CLINICAL TRIAL: NCT01561872
Title: Assessment of an Automated Telesurveillance System on Serious Falls Prevention in an Elderly Suffering From Dementia Specialized Care Unit: the URCC. GET-BETTER Study (Geriatric Environmental Telecare - Behavioral Engineering Technology To Enhance Rehabilitation)
Brief Title: Assessment of an Automated Telesurveillance System on Serious Falls Prevention in an Elderly Suffering From Dementia Specialized Care Unit: the URCC
Acronym: GET-BETTER
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I11 005
Record Dates: First submitted 2012-03-21; First posted 2012-03-23 (Estimated); Last update posted 2015-02-13 (Estimated); Status verified 2015-02

CONDITIONS: Mentally Ill Old Subjects

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- intervention group: Rooms of the patient of the "intervention group" will be equipped of cameras
- reference group: Patient in the "non-equipped" group will have usual care

SUMMARY:
2 URCC in the Limousin region will be equipped with the automated telesurveillance system. Patient will be selected by ward's geriatrician and randomized into two groups after informed consent. One group will have cameras installed and the other will not and will act as a comparison group. Patient will be assessed twice during the study, at admission in (inclusion visit) and at outcome from the URCC (end of study visit). Each assessment implies a standard geriatric assessment, a fall questionnaire, a Neuropsychiatric inventory for behavioral disturbances and a quality of life questionnaire (EQ5D). Every fall will be considered as adverse events and will therefore be listed along the study and characterized in types and number.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged more than 65 years old
* Patient admitted in Limoges or Brive's URCC
* Patient informed consent and/or proxy consent
* Patient covered by the French health insurance

Exclusion Criteria:

* Patient without national health insurance coverage
* Patient with a short term prognosis pathology

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: demented old subjects
Sampling Method: Probability Sample
Enrollment: 350 (Actual)
Dates: Start 2012-04; Primary Completion 2014-11 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
The impact of the automated telesurveillance system | 6 months
  The impact of the automated telesurveillance system on the incidence rate of falls with serious outcomes between the two groups during their hospitalization in URCC.

SECONDARY OUTCOMES:
The impact of the system on the global rate of falls | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Thierry DANTOINE, MD, Study Director — University Hospital, Limoges
Locations (1):
- Limoges University Hospital, Limoges, France